CLINICAL TRIAL: NCT04788641
Title: A Two-Cohort, Randomised Sequence, Cross-over, Open-label Study to Assess the Effect of a Single Dose of Sodium Zirconium Cyclosilicate (SZC) on the Pharmacokinetics of Tacrolimus and Cyclosporin in Healthy Subjects
Brief Title: Study to Assess the Effect of Sodium Zirconium Cyclosilicate on the Pharmacokinetics of Tacrolimus and Cyclosporin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9480C00012; 2020-000515-68 (EudraCT Number)
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hyperkalaemia
Keywords: Pharmacokinetics; Sodium Zirconium Cyclosilicate; Tacrolimus; Cyclosporin; Drug-drug interaction study
MeSH Terms: conditions — Hyperkalemia | interventions — Tacrolimus; Cyclosporine; sodium zirconium cyclosilicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Subjects in Cohort 1 will be randomised in a 1:1 ratio to receive one of the 2 treatment sequences and then cross-over to the other: tacrolimus alone (treatment A) followed by the combination treatment of tacrolimus and SZC (treatment B) or vice versa.
  Interventions: Drug: Tacrolimus; Drug: Sodium Zirconium Cyclosilicate
- Cohort 2 (Experimental): Subjects in Cohort 2 will be randomised in a 1:1 ratio to receive one of the 2 treatment sequences and then cross-over to the other: cyclosporin alone (treatment C) followed by the combination treatment of cyclosporin and SZC (treatment D) or vice versa.
  Interventions: Drug: Cyclosporin; Drug: Sodium Zirconium Cyclosilicate

INTERVENTIONS:
Drug: Tacrolimus — Each subject in this cohort will receive a single dose of oral capsules of tacrolimus on 2 occasions, once alone and once in combination with oral suspension of SZC. Drug administrations will occur after a 12 hour overnight fast.
  Arms: Cohort 1
Drug: Cyclosporin — Each subject will receive a single dose of oral capsules of cyclosporin on 2 occasions, once alone and once in combination with oral suspension of SZC. Drug administrations will occur after a 12 hour overnight fast.
  Arms: Cohort 2
Drug: Sodium Zirconium Cyclosilicate — Each subject will receive single oral doses of SZC with tacrolimus (cohort 1) or cyclosporin (cohort 2) under fasted conditions. The doses will be administered after an overnight fast of at least 12 hours.

SUMMARY:
This study will be an open-label, randomised sequence, 2-period, 2-cohort, 2-treatment in each cohort, cross-over study in healthy subjects (males and females of non-childbearing potential), performed at a single study centre.

DETAILED DESCRIPTION:
The study will comprise:

* A screening period of maximum 28 days;
* Two treatment periods:

  * Treatment Period 1 starts with admission to the Clinical Unit on Day -1, followed by dosing on Day 1 with the assigned treatment (A, B, C, or D) as per assigned cohort and treatment sequence, followed by a washout period of at least 14 days.
  * Treatment Period 2 starts with admission to Clinical Unit on Day -1, followed by dosing on Day 1 with cross-over treatment as per assigned cohort, followed by a follow-up period of 7 to 10 days.
* A follow-up visit/early termination visit at 7 to 10 days after the last investigation medicinal product (IMP) administration.

Subjects will be assigned to either Cohort 1 (tacrolimus) or to Cohort 2 (cyclosporin). Each cohort will have 2 treatment periods. Subjects in each cohort will be randomly assigned to one of 2 treatment sequences (AB|BA or CD|DC) where,

* Treatment A: Tacrolimus
* Treatment B: Tacrolimus + SZC
* Treatment C: Cyclosporin
* Treatment D: Cyclosporin + SZC

ELIGIBILITY:
Inclusion Criteria:

• Healthy male and female subjects aged 18 to 50 years (both inclusive)

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important abnormalities in rhythm, conduction or morphology of the 12-lead safety electrocardiogram (ECG), at screening visit and/or admission to the Clinical Unit.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to SZC, tacrolimus, or cyclosporin.
* Subjects who have previously received SZC.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Koernicke, Dr, Principal Investigator — Parexel Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00012&attachmentIdentifier=4d4be293-ce6b-4b10-abe0-79328caf0fa9&fileName=D9480C00012_Protocol_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00012&attachmentIdentifier=bd271d54-85fe-4919-bb43-2ca84157a0f4&fileName=D9480C00012_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single study centre (Berlin, Germany) between 30 March 2021 to 16 September 2021.
Pre-assignment Details: Participants who met all the inclusion and none of the exclusion criteria were randomized at single center. The screening period was from Day -28 to Day -2. All participants signed and dated the Informed consent form before any study procedures were performed. All the study assessments were performed as per the schedule of assessment.
Groups:
- Cohort 1 (Tacrolimus): Treatment A, Then Treatment B: Participants received a single dose of oral capsules of Tacrolimus on 2 occasions once alone (Treatment A: Tacrolimus) in Treatment Period 1 on Day 1 and once in combination with oral suspension of SZC (Treatment B: Tacrolimus+ SZC) in Treatment Period 2 on Day 1 separated by at least 14 days. Participants had a follow-up period of 7 to 10 days.
- Cohort 1 (Tacrolimus): Treatment B, Then Treatment A: Participants received a single dose of oral capsules of Tacrolimus on 2 occasions once in combination with oral suspension of SZC (Treatment B: Tacrolimus + SZC) in Treatment Period 2 on Day 1 and once alone (Treatment A: Tacrolimus) in Treatment Period 1 on Day 1 and separated by at least 14 days. Participants had a follow-up period of 7 to 10 days.
- Cohort 2 (Cyclosporin): Treatment C, Then Treatment D: Participants received a single dose of oral capsules of Cyclosporin on 2 occasions once alone (Treatment C: Cyclosporin) in Treatment Period 1 on Day 1 and once in combination with oral suspension of SZC (Treatment D: Cyclosporin + SZC) in Treatment Period 2 on Day 1 separated by at least 14 days. Participants had a follow-up period of 7 to 10 days.
- Cohort 2 (Cyclosporin): Treatment D, Then Treatment C: Participants received a single dose of oral capsules of Cyclosporin on 2 occasions once in combination with oral suspension of SZC (Treatment D: Cyclosporin + SZC) in Treatment Period 2 on Day 1 and once alone (Treatment C: Cyclosporin) in Treatment Period 1 on Day 1 and separated by at least 14 days. Participants had a follow-up period of 7 to 10 days.
Period: Treatment Period 1 (4 Days)
Arm/Group | Cohort 1 (Tacrolimus): Treatment A, Then Treatment B | Cohort 1 (Tacrolimus): Treatment B, Then Treatment A | Cohort 2 (Cyclosporin): Treatment C, Then Treatment D | Cohort 2 (Cyclosporin): Treatment D, Then Treatment C
Started | 16 | 15 | 16 | 15
Completed | 16 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (14 Days)
Arm/Group | Cohort 1 (Tacrolimus): Treatment A, Then Treatment B | Cohort 1 (Tacrolimus): Treatment B, Then Treatment A | Cohort 2 (Cyclosporin): Treatment C, Then Treatment D | Cohort 2 (Cyclosporin): Treatment D, Then Treatment C
Started | 16 | 15 | 16 | 15
Completed | 16 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (4 Days)
Arm/Group | Cohort 1 (Tacrolimus): Treatment A, Then Treatment B | Cohort 1 (Tacrolimus): Treatment B, Then Treatment A | Cohort 2 (Cyclosporin): Treatment C, Then Treatment D | Cohort 2 (Cyclosporin): Treatment D, Then Treatment C
Started | 16 | 15 | 16 | 15
Completed | 15 | 15 | 14 | 15
Not Completed | 1 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Participant decided to discontinue further participation | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The randomised set consisted of all participants randomised into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Tacrolimus): Treatment A, Then Treatment B | Cohort 1 (Tacrolimus): Treatment B, Then Treatment A | Cohort 2 (Cyclosporin): Treatment C, Then Treatment D | Cohort 2 (Cyclosporin): Treatment D, Then Treatment C | Total
Number analyzed (Participants) | 16 | 15 | 16 | 15 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The randomised set consisted of all participants randomised into the study.
  Here, the separate rows were created to capture the total Mean(SD) data for each cohort.
  years
    Cohort 1 (Tacrolimus): number analyzed (Participants) | 16 | 15 | 0 | 0 | 31
    Cohort 1 (Tacrolimus) | 38.3 (8.9) | 37.1 (9.6) |  |  | 37.7 (9.1)
    Cohort 2 (Cyclosporin): number analyzed (Participants) | 0 | 0 | 16 | 15 | 31
    Cohort 2 (Cyclosporin) |  |  | 33.2 (9.0) | 30.9 (8.3) | 32.1 (8.6)
Age, Customized [Count of Participants; unit: Participants]
  18 - 50 years | 16 | 15 | 16 | 15 | 62
  51 years and older | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 3
  Male | 15 | 13 | 16 | 15 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 15 | 12 | 13 | 54
  Black or African American | 0 | 0 | 2 | 0 | 2
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Other | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 15 | 15 | 15 | 61

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax)
Description: Effect of co-administered SZC on the Cmax of tacrolimus and cyclosporin in healthy participants was determined.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose of tacrolimus or cyclosporin
Population: The PK analysis set consisted of all participants in the safety analysis set and who had at least 1 quantifiable whole blood concentration post-dose for tacrolimus (Cohort 1) or for cyclosporin (Cohort 2) and who had no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter (pg/ml)
Groups:
- Treatment A: Tacrolimus (5 mg): Participants received a single dose of oral capsules of Tacrolimus.
- Treatment B: Tacrolimus (5 mg) and SZC (15 g): Participants received a single dose of oral capsules of Tacrolimus in combination with oral suspension of SZC.
- Treatment C: Cyclosporin (100 mg): Participants received a single dose of oral capsules of Cyclosporin.
- Treatment D: Cyclosporin (100 mg) and SZC (15 g): Participants received a single dose of oral capsules of Cyclosporin in combination with oral suspension of SZC.
Arm/Group | Treatment A: Tacrolimus (5 mg) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) | Treatment C: Cyclosporin (100 mg) | Treatment D: Cyclosporin (100 mg) and SZC (15 g)
Number analyzed (Participants) | 31 | 30 | 31 | 29
Picogram/milliliter (pg/ml) | 27140 (37.61) | 19350 (35.88) | 593.6 (19.54) | 608.1 (25.28)
Statistical Analysis 1: Comparison: Treatment A: Tacrolimus (5 mg) vs Treatment B: Tacrolimus (5 mg) and SZC (15 g); Tacrolimus; Test type: Other; Geometric LS Mean Ratio (%) = 71.10, 90% CI 2-sided [65.44 to 77.24] — Result based on a mixed effect following a natural logarithmic transformation of the individual PK parameters, with period, treatment, and sequence as fixed effects, and participant nested within sequence as random effects
Statistical Analysis 2: Comparison: Treatment C: Cyclosporin (100 mg) vs Treatment D: Cyclosporin (100 mg) and SZC (15 g); Cyclosporin; Test type: Other; Geometric LS Mean Ratio (%) = 102.9, 90% CI 2-sided [96.11 to 110.1] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: Effect of co-administered SZC on the AUCinf of tacrolimus and cyclosporin in healthy participants was determined.
Time Frame: as for outcome 1
Population: The PK analysis set consisted of all participants in the safety analysis set and who had at least 1 quantifiable whole blood concentration post-dose for tacrolimus (Cohort 1) or for cyclosporin (Cohort 2) and who had no major protocol deviations thought to impact on the analysis of the PK data.
  Here, overall number of participants analyzed are the participants with available data that were analyzed for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram.hour/milliliter
Arm/Group | Treatment A: Tacrolimus (5 mg) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) | Treatment C: Cyclosporin (100 mg) | Treatment D: Cyclosporin (100 mg) and SZC (15 g)
Number analyzed (Participants) | 26 | 27 | 31 | 29
Picogram.hour/milliliter | 267900 (50.20) | 171700 (48.95) | 1884 (25.90) | 1810 (23.91)
Statistical Analysis 1: Comparison: Treatment A: Tacrolimus (5 mg) vs Treatment B: Tacrolimus (5 mg) and SZC (15 g); Tacrolimus; Test type: Other; Geometric LS Mean Ratio (%) = 62.91, 90% CI 2-sided [55.64 to 71.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment C: Cyclosporin (100 mg) vs Treatment D: Cyclosporin (100 mg) and SZC (15 g); Cyclosporin; Test type: Other; Geometric LS Mean Ratio (%) = 97.23, 90% CI 2-sided [92.93 to 101.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast)
Description: Effect of co-administered SZC on the AUClast of tacrolimus and cyclosporin in healthy participants was determined.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram.hour/milliliter
Arm/Group | Treatment A: Tacrolimus (5 mg) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) | Treatment C: Cyclosporin (100 mg) | Treatment D: Cyclosporin (100 mg) and SZC (15 g)
Number analyzed (Participants) | 31 | 30 | 31 | 29
Picogram.hour/milliliter | 240800 (50.79) | 159000 (51.13) | 1792 (26.46) | 1718 (24.39)
Statistical Analysis 1: Comparison: Treatment A: Tacrolimus (5 mg) vs Treatment B: Tacrolimus (5 mg) and SZC (15 g); Tacrolimus; Test type: Other; Geometric LS Mean Ratio (%) = 65.57, 90% CI 2-sided [58.69 to 73.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment C: Cyclosporin (100 mg) vs Treatment D: Cyclosporin (100 mg) and SZC (15 g); Cyclosporin; Test type: Other; Geometric LS Mean Ratio (%) = 97.04, 90% CI 2-sided [92.70 to 101.6] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Reach Maximum Observed Concentration Following Drug Administration (Tmax)
Description: Effect of co-administered SZC on the tmax of tacrolimus and cyclosporin in healthy participants was determined.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A: Tacrolimus (5 mg) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) | Treatment C: Cyclosporin (100 mg) | Treatment D: Cyclosporin (100 mg) and SZC (15 g)
Number analyzed (Participants) | 31 | 30 | 31 | 29
hour | 1.75 [1.00 to 3.00] | 1.50 [0.75 to 3.00] | 1.50 [0.75 to 2.50] | 1.25 [0.98 to 2.52]
Statistical Analysis 1: Comparison: Treatment A: Tacrolimus (5 mg) vs Treatment B: Tacrolimus (5 mg) and SZC (15 g); Tacrolimus; Test type: Other; Geometric LS Mean Ratio (%) = 83.86, 90% CI 2-sided [73.38 to 95.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment C: Cyclosporin (100 mg) vs Treatment D: Cyclosporin (100 mg) and SZC (15 g); Cyclosporin; Test type: Other; Geometric LS Mean Ratio (%) = 97.55, 90% CI 2-sided [87.16 to 109.2] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz)
Description: Effect of co-administered SZC on the t½λz of tacrolimus and cyclosporin in healthy participants was determined.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment A: Tacrolimus (5 mg) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) | Treatment C: Cyclosporin (100 mg) | Treatment D: Cyclosporin (100 mg) and SZC (15 g)
Number analyzed (Participants) | 31 | 30 | 31 | 29
hour | 33.59 (18.72) | 33.31 (22.27) | 9.223 (32.78) | 8.647 (31.12)
Statistical Analysis 1: Comparison: Treatment A: Tacrolimus (5 mg) vs Treatment B: Tacrolimus (5 mg) and SZC (15 g); Tacrolimus; Test type: Other; Geometric LS Mean Ratio (%) = 98.42, 90% CI 2-sided [94.62 to 102.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment C: Cyclosporin (100 mg) vs Treatment D: Cyclosporin (100 mg) and SZC (15 g); Cyclosporin; Test type: Other; Geometric LS Mean Ratio (%) = 94.12, 90% CI 2-sided [85.74 to 103.3] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs
Description: Safety and tolerability of co-administration of SZC and tacrolimus/cyclosporin as compared to tacrolimus/cyclosporin alone was assessed.
Time Frame: From the time of IMP administration (Day 1) to Follow-up/Early Termination Visit (7-10 days after last IMP administration) [up to 4 weeks]
Population: All participants who received at least 1 dose of IMP were included in the safety analysis for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Tacrolimus (5 mg) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) | Treatment C: Cyclosporin (100 mg) | Treatment D: Cyclosporin (100 mg) and SZC (15 g)
Number analyzed (Participants) | 31 | 30 | 31 | 29
Participants
  Any AE | 7 | 13 | 8 | 7
  Any AE with outcome = death | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of IMP | 0 | 0 | 1 | 0
  Any AE leading to withdrawal from study | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the time of IMP administration (Day 1) to Follow-up/Early Termination Visit (7-10 days after last IMP administration) [up to 4 weeks]
Arm/Group | Treatment A: Tacrolimus (5 mg) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) | Treatment C: Cyclosporin (100 mg) | Treatment D: Cyclosporin (100 mg) and SZC (15 g)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 7/31 | 13/30 | 8/31 | 7/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Tacrolimus (5 mg) (N=31) | Treatment B: Tacrolimus (5 mg) and SZC (15 g) (N=30) | Treatment C: Cyclosporin (100 mg) (N=31) | Treatment D: Cyclosporin (100 mg) and SZC (15 g) (N=29)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (2)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT04788641/Prot_SAP_000.pdf